CLINICAL TRIAL: NCT00177853
Title: A Phase I Study of Celecoxib, Irinotecan and Concurrent Radiotherapy in the Preoperative Treatment of Pancreatic Cancer
Brief Title: Celecoxib, Irinotecan and Concurrent Radiotherapy in Preoperative Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: terminated
Sponsor: University of Pittsburgh (Other)
Collaborators: Pharmacia and Upjohn (Industry)
Responsible Party: A. James Moser, MD, UPCI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-128
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced pancreatic cancer; invasion of major arteries and veins around pancreas; No prior radiation or chemo
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Celecoxib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Celecoxib, Irinotecan and Concurrent Radiotherapy
  Interventions: Drug: celecoxib; Drug: irinotecan; Procedure: concurrent radiotherapy

INTERVENTIONS:
Drug: celecoxib — Patients will start celecoxib (200mg PO BID) beginning 3-5 days prior to chemoradiation at home and receive the drug until 30 days following the completion of chemoradiation.
  Other Names: Celebrex
Drug: irinotecan — Preoperative chemoradiation will consist of escalating doses of irinotecan (30 50 mg/m2 IV) once weekly for a total of 4 doses.
  Other Names: Camptosar
Procedure: concurrent radiotherapy — 50.4 cGy of standard external beam radiation. The radiation will be given in 28 treatments of 1.8 cGy per treatment over 5.5 weeks. This will be given in an outpatient setting.

SUMMARY:
The purposes of this study are to examine the effects of a new combination of drugs, celecoxib (Celebrex®) and irinotecan (CPT-11), with standard radiation therapy on people before they undergo surgery; to determine what effects this combination has on pancreatic cancer; and to determine the highest dose of celecoxib and irinotecan that can be given safely without causing severe side effects. While not an endpoint, it is hoped that this combination will also shrink tumors enough for excision.

DETAILED DESCRIPTION:
The purposes of this study are to examine the effects of a new combination of drugs, celecoxib (Celebrex®) and irinotecan (CPT-11), with standard radiation therapy on people before they undergo surgery; to determine what effects this combination has on pancreatic cancer; and to determine the highest dose of celecoxib and irinotecan that can be given safely without causing severe side effects. While not an endpoint, it is hoped that this combination will also shrink tumors enough for excision.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced carcinoma of the pancreas
* Arterial invasion or encasement
* Invasion/encasement of the portomesenteric veins
* Patients who have been previously denied operation
* Obstructive jaundice must be drained with a polyethylene biliary stent or surgical bypass prior to beginning treatment.
* White blood cell count > 3500 per ml and platelet count > 100,000 per ml
* Serum creatinine ≤ 1.5 mg/dl
* Bilirubin ≤ 1.5
* ECOG performance status < 2

Exclusion Criteria:

* Prior chemotherapy, radiotherapy, or investigational agents for pancreatic cancer
* Evidence of distant metastasis or malignant lymphadenopathy
* Concurrent malignancies
* History of allergic reactions to celecoxib or to sulfa drugs
* No non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, magnesium or aluminum containing antacids, fluconazole or lithium may be administered within 5 days of study entry, during the study and for the 30 days following the completion of all study treatments.
* Pregnant women and lactating women
* Uncontrolled or serious intercurrent illness
* HIV-positive patients receiving combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine efficacy of combination of irinotecan, celecoxib and concurrent radiotherapy on pancreatic cancer; determine highest/safest doses of these drugs | 12 weeks

SECONDARY OUTCOMES:
Tumor diminishment for safe excision | 75 days

CONTACTS AND LOCATIONS:
Overall Officials: A. J. Moser, MD, Principal Investigator — University of Pittsburgh Medical Center Department of Surgery, Division of Surgical Oncology
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States